CLINICAL TRIAL: NCT02417727
Title: A Feasibility Study of Deep Brain Recordings for Learning and Memory
Brief Title: Feasibility Study of Deep Brain Recordings for Learning and Memory
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150102; 15-N-0102
Record Dates: First submitted 2015-04-15; First posted 2015-04-16 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2015-10-23

CONDITIONS: Movement Disorders
Keywords: MEMORY TESTING; Biomarkers; Learning
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Some people with movement disorders are in another NIH protocol. They will have electrodes placed in deep brain areas. They may do tasks before, during, and after surgery. Researchers want to learn more about how brain cells and networks work while people learn and remember. They want to use the data from the other NIH study to do this.

Objective:

- To share data from before and during deep brain stimulation surgery. The data will be used in a study of how the brain learns and remembers.

Eligibility:

- People at least 18 years old who are in protocol 11-N-0211 and have certain movement disorders.

Design:

* As part of protocol 11-N-0211, data on participants brainwave activity is collected. In this protocol, they will have that data stored and shared.
* Researchers will access imaging data from deep brain stimulation surgery.
* Researchers will access other medical records.

DETAILED DESCRIPTION:
OBJECTIVES:

The purpose of this protocol is to share neural data collected before and during deep brain stimulation surgery with the University of Pennsylvania to identify biomarkers of successful learning and memory.

STUDY POPULATION:

Up to twenty (20) adult subjects who are participating in NIH protocol 11-N-0211 Deep Brain Stimulation Surgery for Movement Disorders who provide written informed consent for sharing and the additional use of their data.

STUDY DESIGN:

This protocol only involves providing consent to share learning and memory data collected under Protocol 11-N-0211. There are no separate or additional participant procedures involved in this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults at least age 18

Currently enrolled in 11-N-0211

EXCLUSION CRITERIA:

Unable to provide own informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-23; Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Permission to share data from partiicpation on NIH protocol #11-N-0211 | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)